CLINICAL TRIAL: NCT06381466
Title: A Phase I, Randomized, Single Blinded, Placebo-controlled Study to Assess the Safety, Tolerability, and Pharmacokinetics of AZD0233 Following Single and Multiple Ascending Dose Administration in Healthy Male and Female Participants 18 to 50 Years of Age.
Brief Title: A Study to Investigate Safety, Tolerability, and Pharmacokinetics of Oral AZD0233 Compared With Placebo in Healthy Adult Participants.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study has been terminated due to adverse finding in a non-clinical, chronic toxicology study.
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: D7250C00001
Record Dates: First submitted 2024-03-29; First posted 2024-04-24 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Dilated Cardiomyopathy
Keywords: Heart failure; Single Ascending Dose (SAD); Multiple Ascending Dose (MAD); Pharmacokinetics
MeSH Terms: conditions — Cardiomyopathy, Dilated; Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Part A (SAD): Cohort 1A - AZD0233 (dose 1) (Experimental): Healthy participants will receive AZD0233 (dose 1) orally as a single ascending dose.
  Interventions: Drug: AZD0233
- Part A (SAD): Cohort 2A - AZD0233 (dose 2) (Experimental): Healthy participants will receive AZD0233 (dose 2) orally as a single ascending dose.
  Interventions: Drug: AZD0233
- Part A (SAD): Cohort 3A - AZD0233 (dose 3) (Experimental): Healthy participants will receive AZD0233 (dose 3) orally as a single ascending dose.
  Interventions: Drug: AZD0233
- Part A (SAD): Cohort 4A - AZD0233 (dose 4) (Experimental): Healthy participants will receive AZD0233 (dose 4) orally as a single ascending dose.
  Interventions: Drug: AZD0233
- Part A (SAD): Cohort 5A - AZD0233 (dose 5) (Experimental): Healthy participants will receive AZD0233 (dose 5) orally as a single ascending dose.
  Interventions: Drug: AZD0233
- Part B (MAD): Cohort 1B - AZD0233 (dose 6) (Experimental): Healthy participants will receive AZD0233 (dose 6) orally as a multiple ascending dose.
  Interventions: Drug: AZD0233
- Part B (MAD): Cohort 2B - AZD0233 (dose 7) (Experimental): Healthy participants will receive AZD0233 (dose 7) orally as a multiple ascending dose.
  Interventions: Drug: AZD0233
- Part B (MAD): Cohort 3B - AZD0233 (dose 8) (Experimental): Healthy participants will receive AZD0233 (dose 8) orally as a multiple ascending dose.
  Interventions: Drug: AZD0233
- Part A (SAD): Placebo cohort (Placebo Comparator): Healthy participants will receive placebo orally as a single ascending dose.
  Interventions: Drug: AZD0233 Placebo
- Part B (MAD): Placebo cohort (Placebo Comparator): Healthy participants will receive placebo orally as a multiple ascending dose.
  Interventions: Drug: AZD0233 Placebo
- Part A (SAD): Food Effect (FE) extended Cohort 3A (Experimental): Healthy participants from Cohort 3A will participate in this extended cohort after a washout period of 24 hours.
  Interventions: Drug: AZD0233

INTERVENTIONS:
Drug: AZD0233 — Randomized participants will receive AZD0233 orally as a single ascending dose (dose 1, dose 2, dose 3, dose 4 or dose 5) or multiple ascending dose (dose 6, dose 7 or dose 8)
  Arms: Part A (SAD): Cohort 1A - AZD0233 (dose 1); Part A (SAD): Cohort 2A - AZD0233 (dose 2); Part A (SAD): Cohort 3A - AZD0233 (dose 3); Part A (SAD): Cohort 4A - AZD0233 (dose 4); Part A (SAD): Cohort 5A - AZD0233 (dose 5); Part A (SAD): Food Effect (FE) extended Cohort 3A; Part B (MAD): Cohort 1B - AZD0233 (dose 6); Part B (MAD): Cohort 2B - AZD0233 (dose 7); Part B (MAD): Cohort 3B - AZD0233 (dose 8)
Drug: AZD0233 Placebo — Randomized participants will receive matching placebo orally as a SAD or MAD.
  Other Names: Placebo
  Arms: Part A (SAD): Placebo cohort; Part B (MAD): Placebo cohort

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and pharmacokinetics of AZD0233 following single and multiple ascending dose (SAD and MAD) administration in healthy participants.

DETAILED DESCRIPTION:
This is a Phase I, first time in human, single-blinded, randomized, placebo-controlled study in healthy adult male and female (of non-childbearing potential) participants performed at a single Clinical Unit.

The study will be carried out in 2 parts: Part A and Part B. Eight participants will participate in each cohort. Within each cohort, 6 participants will be randomized to receive AZD0233, and 2 participants will be randomized to receive placebo.

Part A of the study will be a sequential SAD design. Five dose levels of AZD0233 are planned to be investigated (dose 1 to dose 5), 2 (dose 3 and dose 4) of which will also be assessed in participants of Japanese descent.

Part A of the study will comprise:

* A Screening Period of maximum 26 days (Day -28 to Day -2).
* An inpatient Period of up to 7 days (Day -1 to Day 6):

  * Cohorts 1A, 2A, 3A (Japanese sub-Cohort only), 4A (including a Japanese sub-Cohort), and 5A: participants will be resident at the Clinical Unit from Day -1 before study intervention administration until Day 4 (72 hours after administration of the study intervention).
  * Cohort 3A [food effect (FE)]: Participants will be resident at the Clinical Unit from Day -1 before study intervention administration and will check-out on Day 6 (72 hours after administration of the study intervention). The impact of food intake on the PK of AZD0233 will be evaluated in the same participants in Cohort 3A after a 24-hour washout period on Day 2.

Note: Japanese sub-Cohort from Cohort 3A will not be part of the FE study.

• A Follow-up Period of 7 days after the administration of the study intervention which will consist of 1 Follow-up Visit on Day 8 for Cohorts 1A, 2A, 3A (Japanese sub-Cohort only), 4A (including a Japanese sub-Cohort), and 5A and one Follow-up Visit on Day 10 for Cohort 3A, for which participants will return to the Clinical Unit for follow-up assessments.

Part B will be a sequential MAD study. Participants will be naïve to AZD0233, i.e., will not have participated in Part A of this study. There will be 3 dose levels in 4 cohorts, including a sub-cohort of participants of Japanese descent at the highest dose.

Part B will consist of:

* A Screening Period of maximum 26 days (Day -28 to Day -2).
* An Inpatient Period of 14 days (Day -1 to Day 13): Participants will be resident at the Clinical Unit from Day -1 before study intervention administration until Day 13 (>48 hours after administration of the last dose of study intervention in case of QD (once daily) dosing and >36 hours after the last dose for BID (twice a day) in case of dosing).
* A Follow-up Period of 7 days after the administration of the last dose of study intervention which will consist of 2 Follow-up Visits on Day 15 and Day 17.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female participants with suitable veins for cannulation or repeated venipuncture.
* All females must have a negative pregnancy test at the Screening Visit and on admission to the Clinical Unit.
* Females of non-childbearing potential must be confirmed at the Screening Visit by fulfilling one of the following criteria:

  1. Post-menopausal defined as amenorrhea for at least 12 months following cessation of all exogenous hormonal treatments and follicle-stimulating hormone (FSH) levels in the post-menopausal range.
  2. Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy but not tubal ligation.
* Sexually active fertile male participants with partners of childbearing potential must adhere to the specified contraception methods from the time of first administration of study intervention until 3 months after the study Follow-up Visit.
* Have a body mass index between 18 and 30 kg/m² inclusive and weigh at least 50 kg.

Note: For Japanese sub-Cohort minimum weight of 45 kg is acceptable.

• For the healthy Japanese sub-Cohorts: healthy Japanese participants (e.g., natives of Japan or Japanese Americans) are defined as having both parents and 4 grandparents who are Japanese. This includes healthy second and third generation participants of Japanese descent whose parents or grandparents are living in a country other than Japan.

Exclusion Criteria:

* History of any clinically important disease or disorder which may either put the participant at risk because of participation in the study or influence the results or the participant's ability to participate in the study.
* History or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of study intervention.
* Any clinically important abnormalities in clinical chemistry, hematology, urinalysis, laboratory values or vital signs at Screening and/or first admission to the Clinical Unit.
* Any clinically important abnormalities in rhythm, conduction or morphology of the resting electrocardiogram (ECG) and any clinically important abnormalities in the 12-lead ECG that may interfere with the interpretation of corrected QT (QTc) interval changes in heart rate.
* Current smokers or those who have smoked or used nicotine products (including e-cigarettes) within the previous 3 months prior to Screening.
* Known or suspected history of alcohol or drug abuse or excessive intake of alcohol.
* Positive screen for drugs of abuse, or alcohol or cotinine at Screening or on each admission to the Clinical Unit.
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, or history of hypersensitivity to drugs of a similar class to AZD0233.
* Use of drugs with enzyme [Cytochrome P450 3A (CYP3A)]/ transporter [breast cancer resistance protein (BCRP) and organic anion transporting polypeptide 1B (OATP1B)] inducing/ inhibiting properties such as St John's Wort within 3 weeks prior to the first administration of study intervention.
* Use of any prescribed or nonprescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, mega dose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of study intervention or longer if the medication has a long half-life. Hormone replacement therapy medications are allowed for female participants.
* Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 30 days or 5 half-lives (whichever is longest) of the first administration of investigational medicinal product (IMP) in this study. The period of exclusion begins one month after the final dose.
* Participants who have previously received AZD0233.
* Active systemic bacterial, viral, or fungal infection within 14 days prior to dosing or presence of fever (confirmed tympanic body temperature > 37.6 °C) within 14 days prior to dosing on Day 1 depending on experienced symptoms.
* Clinically significant serious active and chronic infections within 60 days prior to randomization.
* Known history of primary immunodeficiency (congenital or acquired) or an underlying condition that predisposes to infection.
* Concomitant immunosuppressive and/or steroid treatment.
* Any positive result on Screening for serum hepatitis B surface antigen (HBsAg), hepatitis B core antibody (anti-HBc), hepatitis C antibody, human immunodeficiency virus (HIV).
* Clinical signs and symptoms consistent with COVID-19.
* Participants who are vegans or have medical dietary restrictions.
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the Clinical Unit).
* Judgment by the investigator that the participant should not participate in the study if they have any ongoing or recent (ie, during the Screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.
* Participants who cannot communicate reliably with the investigator.
* Vulnerable participants, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) and serious adverse events (SAEs) | From screening (Day -28) to follow-up visit (Day 17)
  To assess the safety and tolerability of AZD0233 following oral administration of single ascending doses (Part A) and multiple ascending doses (Part B) and to estimate the maximum tolerated dose (if within pre-defined exposure limits).

SECONDARY OUTCOMES:
Maximum observed plasma (peak) drug concentration (Cmax) of AZD0233 | Day 1 (Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 16 hours), Day 2 (24 hours and 36 hours post-dose) and Day 3 (48 hours post-dose)
  To characterize the single-dose and steady state pharmacokinetics (PK) of AZD0233 following oral administration of AZD0233 and to assess the impact of food on the single-dose PK of AZD0233 (Dose 3 FE extended cohort in Cohort 3A of Part A).
Area under the plasma concentration-curve from zero to the last quantifiable concentration (AUClast) of AZD0233 | Day 1 (Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 16 hours), Day 2 (24 hours and 36 hours post-dose) and Day 3 (48 hours post-dose)
  To characterize the single-dose and steady state PK of AZD0233 following oral administration of AZD0233 and to assess the impact of food on the single-dose PK of AZD0233 (Dose 3 FE extended cohort in Cohort 3A of Part A).
Area under the concentration-time curve in the dose interval (AUCtau) of AZD0233 | Day 1 (Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 16 hours), Day 2 (24 hours and 36 hours post-dose) and Day 3 (48 hours post-dose)
  To characterize the single-dose and steady state PK of AZD0233 following oral administration of AZD0233 and to assess the impact of food on the single-dose PK of AZD0233 (Dose 3 FE extended cohort in Cohort 3A of Part A).
Area under plasma concentration time-curve from zero to infinity (AUCinf) of AZD0233 | Day 1 (Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 16 hours), Day 2 (24 hours and 36 hours post-dose) and Day 3 (48 hours post-dose)
  To characterize the single-dose and steady state PK of AZD0233 following oral administration of AZD0233 and to assess the impact of food on the single-dose PK of AZD0233 (Dose 3 FE extended cohort in Cohort 3A of Part A).
Time to reach peak or maximum observed concentration or response following drug administration (tmax) of AZD0233 | Day 1 (Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 16 hours), Day 2 (24 hours and 36 hours post-dose) and Day 3 (48 hours post-dose)
  To characterize the single-dose and steady state PK of AZD0233 following oral administration of AZD0233 and to assess the impact of food on the single-dose PK of AZD0233 (Dose 3 FE extended cohort in Cohort 3A of Part A).
Terminal elimination half-life (t1/2) of AZD0233 | Day 1 (Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 16 hours), Day 2 (24 hours and 36 hours post-dose) and Day 3 (48 hours post-dose)
  To characterize the single-dose and steady state PK of AZD0233 following oral administration of AZD0233 and to assess the impact of food on the single-dose PK of AZD0233 (Dose 3 FE extended cohort in Cohort 3A of Part A).
Apparent total body clearance of drug from plasma after extravascular administration (CL/F) of AZD0233 | Day 1 (Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 16 hours), Day 2 (24 hours and 36 hours post-dose) and Day 3 (48 hours post-dose)
  To characterize the single-dose and steady state PK of AZD0233 following oral administration of AZD0233 and to assess the impact of food on the single-dose PK of AZD0233 (Dose 3 FE extended cohort in Cohort 3A of Part A).
Apparent volume of distribution at steady state following extravascular administration (Vz/F) of AZD0233 | Day 1 (Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 16 hours), Day 2 (24 hours and 36 hours post-dose) and Day 3 (48 hours post-dose)
  To characterize the single-dose and steady state PK of AZD0233 following oral administration of AZD0233 and to assess the impact of food on the single-dose PK of AZD0233 (Dose 3 FE extended cohort in Cohort 3A of Part A).
Terminal rate constant (λz) of AZD0233 | Day 1 (Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 16 hours), Day 2 (24 hours and 36 hours post-dose) and Day 3 (48 hours post-dose)
  To characterize the single-dose and steady state PK of AZD0233 following oral administration of AZD0233 and to assess the impact of food on the single-dose PK of AZD0233 (Dose 3 FE extended cohort in Cohort 3A of Part A).
Accumulation ratio for Cmax (Rac Cmax) of AZD0233 | Day 1 (Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 16 hours), Day 2 (24 hours and 36 hours post-dose) and Day 3 (48 hours post-dose)
  To characterize the single-dose and steady state PK of AZD0233 following oral administration of AZD0233 and to assess the impact of food on the single-dose PK of AZD0233 (Dose 3 FE extended cohort in Cohort 3A of Part A).
Accumulation ratio for AUC (Rac AUC) of AZD0233 | Day 1 (Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 16 hours), Day 2 (24 hours and 36 hours post-dose) and Day 3 (48 hours post-dose)
  To characterize the single-dose and steady state PK of AZD0233 following oral administration of AZD0233 and to assess the impact of food on the single-dose PK of AZD0233 (Dose 3 FE extended cohort in Cohort 3A of Part A).
Renal clearance (CLR) of AZD0233 | Spot sample at pre-dose and pooled urine at Day 1 (0-3, 3-6, 6-9, 9-12, and 12-24 hours post-dose), Day 2 (24-36 hours post dose) and Day 3 (36-48 hours post-dose).
  To characterize the single-dose and steady state PK of AZD0233 following oral administration of AZD0233 and to assess the impact of food on the single-dose PK of AZD0233 (Dose 3 FE extended cohort in Cohort 3A of Part A).
Cumulative amount of unchanged drug excreted into urine from time t1 to time t2 [Ae(t1-t2)] of AZD0233 | Spot sample at pre-dose and pooled urine at Day 1 (0-3, 3-6, 6-9, 9-12, and 12-24 hours post-dose), Day 2 (24-36 hours post dose) and Day 3 (36-48 hours post-dose).
  To characterize the single-dose and steady state PK of AZD0233 following oral administration of AZD0233 and to assess the impact of food on the single-dose PK of AZD0233 (Dose 3 FE extended cohort in Cohort 3A of Part A).
Percentage of dose excreted unchanged in urine from time t1 to t2 [Fe(t1-t2)] of AZD0233 | Spot sample at pre-dose and pooled urine at Day 1 (0-3, 3-6, 6-9, 9-12, and 12-24 hours post-dose), Day 2 (24-36 hours post dose) and Day 3 (36-48 hours post-dose).
  To characterize the single-dose and steady state PK of AZD0233 following oral administration of AZD0233 and to assess the impact of food on the single-dose PK of AZD0233 (Dose 3 FE extended cohort in Cohort 3A of Part A).

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/